CLINICAL TRIAL: NCT02398227
Title: Treatment of PTSD in Residents of Battered Women's Shelters
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Akron (Other)
Collaborators: Brown University (Other); Summa Health System (Other); Kent State University (Other); Pacific Institute for Research and Evaluation (Other)
Responsible Party: Principal Investigator, Dawn Johnson, Associate Professor, The University of Akron
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01MH095767 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2015-03-25 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: PTSD
Keywords: Battered Women; Trauma; Domestic Violence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HOPE (Experimental): Cognitive Behavioral Treatment Program for PTSD
  Interventions: Behavioral: HOPE
- PCT (Active Comparator): Present Centered Therapy for PTSD
  Interventions: Behavioral: PCT

INTERVENTIONS:
Behavioral: HOPE — Cognitive Behavioral Treatment for PTSD in Battered Women
  Arms: HOPE
Behavioral: PCT — Present Centered Therapy for PTSD
  Arms: PCT

SUMMARY:
This is a study comparing a new treatment (HOPE) to supportive therapy in the treatment of PTSD in residents of battered women's shelters.

DETAILED DESCRIPTION:
Research suggests that approximately 1 in 4 women report a history of intimate partner violence (IPV), and IPV is associated with severe psychological problems, especially PTSD. Battered women's shelters annually provide emergency shelter to approximately 300,000 women and children. A prime time to intervene with IPV victims might be when they enter shelter and have already initiated a change in their life. Standard shelter care typically includes case management to help women access resources that can assist them in establishing long-term safety for themselves and their children. However, PTSD symptoms may compromise victims' ability to effectively use integral community resources, as well as their ability to appropriately react to threat relevant information, interfering with their ability to establish safety for themselves and their children. As such, research has found PTSD to be associated with re-abuse in victims of IPV.

Despite the significant morbidity associated with IPV-related PTSD, our treatment, Helping to Overcome PTSD through Empowerment (HOPE), is the only extant treatment to date that has been developed to specifically target IPV-related PTSD in residents of battered women's shelters. Cognitive-behavioral treatments (CBT) for PTSD have been shown to be effective with multiple populations but do not address the unique needs of recent IPV victims. HOPE, a shelter-based, individual, brief CBT treatment for PTSD in victims of IPV, addresses IPV victims' current needs of safety, self-care, protection, and empowerment, as well as the exchange of information on PTSD symptoms and how these symptoms interfere with the use of shelter and community resources and their ability to establish safety. HOPE was specifically designed to serve as an evidence-based model program that could be implemented in a wide-range of shelter programs across the United States. The current proposal builds on the foundation of our NIMH-funded treatment development study (R34MH080786). Pilot work with HOPE supports the initial acceptability and feasibility of this new treatment. IPV victims who received a significant dose of HOPE were 12 times less likely than women received only standard shelter services to report being re-abused after leaving shelter. Further, women who received HOPE displayed fewer PTSD arousal and avoidance symptoms of PTSD, less depression, and greater social support and empowerment relative to women who did not receive HOPE. The overall aim of this project is to test the efficacy of HOPE relative to supportive therapy (i.e., Present Centered Therapy, PCT) in a sample of 186 female residents of battered women's shelters with IPV-related PTSD. In an effort to facilitate future dissemination of HOPE, sessions will be delivered by community therapists and the study will be conducted in a range of shelter systems. Furthermore, the current proposal, unlike the pilot study, will compare HOPE to an attention matched control condition, have a longer follow-up period, will assess the impact of HOPE on child abuse potential, and will incorporate objective measures of stress responding (e.g., attentional biases and physiological reactivity to trauma cues), explore mediators and moderators of treatment, and evaluate the cost effectiveness of HOPE.

The Specific Aim of this proposal is to conduct a randomized controlled trial comparing HOPE to PCT in residents of battered women shelters with IPV-related PTSD. The study will test the following hypotheses:

Primary Hypotheses: HOPE will be significantly more efficacious than PCT in reducing participants' IPV-related PTSD symptoms and severity of re-abuse over a one-year follow-up.

Secondary Hypotheses: Associated Symptoms, Psychosocial Functioning, and Cost:

* HOPE will be significantly more efficacious than PCT in decreasing participants' depressive symptoms and child abuse potential; in increasing participants' degree of empowerment, quality of life, degree and quality of social support, effective use of resources, and traumatic cognitions over a one-year follow-up.
* Shelter residents who receive HOPE will display reduced biases in attention to threat-related information and normalization of physiological reactivity to trauma cues, relative to women who receive PCT over a one-year follow-up.
* We also plan to evaluate the cost-effectiveness of HOPE measured by cost per quality adjusted life year saved (QULY).

We will also explore the following hypotheses regarding potential mediators and moderators of HOPE:

* The effect HOPE has on PTSD over the one-year follow-up will be mediated by participants' degree of empowerment, effective use of resources, and traumatic cognitions at post-treatment.
* HOPE participants' PTSD symptoms post-treatment will mediate participants' severity of re-abuse over the one-year follow-up period.
* We also plan to explore whether the following baseline variables are moderators of treatment response: minority status, IPV and PTSD severity, attentional biases to threat related information, and physiological reactivity to trauma cues.

HOPE, a novel treatment for battered women with IPV-related PTSD, has the potential to provide a national model of care for a vulnerable, underserved, and understudied population.

ELIGIBILITY:
Inclusion Criteria:

* must be resident in one of the 6 participating shelters,
* IPV in month prior to shelter,
* PTSD

Exclusion Criteria:

* substance dependence in last 3 months,
* change in meds in last month,
* Bipolar d/o,
* psychosis,
* active suicidality

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Johnson, Ph.D., Principal Investigator — The University of Akron
Locations (1):
- University of Akron, Akron, Ohio, United States

REFERENCES:
- [Derived] Gonzalez A, Haws JK, Alshabani N, Zlotnick C, Johnson DM. Cyber abuse and posttraumatic stress disorder among racially diverse women who have resided in domestic violence shelters: A longitudinal approach. Psychol Trauma. 2025 Jun;17(Suppl 1):S105-S114. doi: 10.1037/tra0001868. Epub 2025 Jan 27. PMID 39869706

RESULTS

PARTICIPANT FLOW:
Groups:
- Present Centered Therapy (PCT): Present Centered Therapy for PTSD
  PCT: Present Centered Therapy for PTSD
Period: Overall Study
Arm/Group | HOPE | Present Centered Therapy (PCT)
Started | 83 | 89
Completed | 56 | 71
Not Completed | 27 | 18
Not completed — Lost to Follow-up | 21 | 12
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Removed from treatment and dropped out | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HOPE | Present Centered Therapy (PCT) | Total
Number analyzed (Participants) | 83 | 89 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 89 | 172
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 34.5 [19 to 59] | 36 [19 to 59] | 35.13 [19 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 89 | 172
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 80 | 87 | 167
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 43 | 76
  White | 41 | 39 | 80
  More than one race | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 83 | 89 | 172
Clinician-Administered PTSD Scale (CAPS) [Mean (Standard Deviation); unit: units on a scale] — Clinical Interview assessing symptoms of Posttraumatic Stress Disorder (PTSD) scores can range from 0 to 136 with higher scores reflecting greater PTSD severity
  units on a scale | 72.11 (20.87) | 77.82 (21.12) | 75.06 (21.14)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: Clinical Interview assessing symptoms of Posttraumatic Stress Disorder (PTSD) scores can range from 0 to 136 with higher scores reflecting greater PTSD severity Adjusted means with baseline scores as a covariate are reported
Time Frame: baseline, post-shelter, post-treatment, 6 months post-treatment, 1 year post-treatment
Population: Analysis include those participants who completed each follow-up time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HOPE | Present Centered Therapy (PCT)
Number analyzed (Participants) | 53 | 70
units on a scale
  post-shelter | 48.08 (25.36) | 52.39 (28.05)
  post-treatment | 31.75 (22.47) | 34.43 (28.33)
  6 month post-treatment | 29.36 (28.36) | 32.63 (27.33)
  1 year post-treatment | 27.32 (24.96) | 29.00 (28.03)
Statistical Analysis 1: Comparison: HOPE vs Present Centered Therapy (PCT); Test type: Superiority; p = .968, ANCOVA; p value reported for overall effect across all-time points between treatment arms

2. Primary Outcome: Severity of Violence Against Women Scale (SVAWS)
Description: Severity of Violence Against Women Scale total score. Scores can range from 0 to 138 with higher scores reflecting greater degree of violence/abuse.Adjusted means with baseline scores as a covariate are reported
Time Frame: baseline, post-shelter, post-treatment, 6-month post-treatment, 1 year post-treatment
Population: Analysis only include those who completed all time-points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOPE | Present Centered Therapy (PCT)
Number analyzed (Participants) | 53 | 69
score on a scale
  post-shelter | 7.81 (15.37) | 13.89 (28.74)
  post-treatment | 3.47 (8.82) | 1.10 (3.86)
  6-month post-shelter | 3.42 (13.51) | 2.73 (8.55)
  1-year post-treatment | 2.40 (9.03) | 3.68 (12.88)
Statistical Analysis 1: Comparison: HOPE vs Present Centered Therapy (PCT); Test type: Superiority; p = .560, ANCOVA; p value reported for overall effect across all-time points between treatment arms

ADVERSE EVENTS:
Time Frame: 12-month follow-up.
Description: 12-month follow up.
Arm/Group | HOPE | Present Centered Therapy (PCT)
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/89
Serious Adverse Events (participants affected / at risk) | 56/83 | 56/89
Other Adverse Events (participants affected / at risk) | 75/83 | 76/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HOPE (N=83) | Present Centered Therapy (PCT) (N=89)
Life Threatening Experience or Trauma (Social circumstances) | 28 (58) | 33 (79)
Life Threatening Experience and Sexual Assault (Social circumstances) | 1 (1) | 2 (12)
Significant Clinical Deterioration Suicidality (Psychiatric disorders) | 4 (8) | 1 (1)
Active Homicidality (Psychiatric disorders) | 2 (2) | 0 (0)
Psychiatric Inpatient Hospitalization (Psychiatric disorders) | 10 (13) | 12 (18)
Hospitalization Related to Domestic Violence (Social circumstances) | 2 (3) | 4 (9)
Other Hospitalization (Social circumstances) | 25 (49) | 29 (62)
Receipt of a Serious Health Diagnosis (Social circumstances) | 3 (4) | 4 (4)
Sexual Assault (Social circumstances) | 12 (29) | 9 (21)
Reporting to Children's Services (Social circumstances) | 4 (5) | 6 (8)
Criminal Charge or Arrest (Social circumstances) | 2 (2) | 1 (2)
Persistent or Significant Disability or Impairment (Social circumstances) | 0 (0) | 0 (0)
Pregnancy Complications (Social circumstances) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HOPE (N=83) | Present Centered Therapy (PCT) (N=89)
Non-life Threatening Abuse or Trauma (Social circumstances) | 74 (297) | 73 (280)
Substance Use (Psychiatric disorders) | 12 (16) | 12 (15)
Significant Clinical Deterioration CAPS (Psychiatric disorders) | 1 (1) | 5 (8)
Confidentiality Breach (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-05-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT02398227/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2011-10-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT02398227/Prot_SAP_001.pdf